CLINICAL TRIAL: NCT03844945
Title: A Prospective, Double-masked, Randomized, Multicenter, Placebo-controlled, Parallel-group Study Assessing the Safety, Ocular Hypotensive Efficacy and Optimum Dose Concentration to be Used Clinically of Netarsudil Ophthalmic Solution in Subjects With Open-angle Glaucoma or Ocular Hypertension in Japan
Brief Title: Efficacy and Systemic Safety of Netarsudil 0.01%, 0.02%, 0.04% Relative to Placebo in Subjects With Open-angle Glaucoma or Ocular Hypertension in Japan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AR-13324-CS208
Record Dates: First submitted 2019-02-15; First posted 2019-02-19 (Actual); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
Keywords: Glaucoma; Ocular Hypertension; Open-Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Netarsudil Ophthalmic Solution 0.01% (Experimental): 1 drop daily into each eye in the evening for 28 days
  Interventions: Drug: Netarsudil Ophthalmic Solution 0.01%
- Netarsudil Ophthalmic Solution 0.02% (Experimental): 1 drop daily into each eye in the evening for 28 days
  Interventions: Drug: Netarsudil Ophthalmic Solution 0.02%
- Netarsudil Ophthalmic Solution 0.04% (Experimental): 1 drop daily into each eye in the evening for 28 days
  Interventions: Drug: Netarsudil Ophthalmic Solution 0.04%
- Netarsudil Ophthalmic Solution Placebo (Placebo Comparator): 1 drop daily into each eye in the evening for 28 days
  Interventions: Other: Netarsudil Ophthalmic Solution Placebo

INTERVENTIONS:
Drug: Netarsudil Ophthalmic Solution 0.01% — Topical sterile ophthalmic solution
  Arms: Netarsudil Ophthalmic Solution 0.01%
Drug: Netarsudil Ophthalmic Solution 0.02% — Topical sterile ophthalmic solution
  Other Names: Rhopressa®
  Arms: Netarsudil Ophthalmic Solution 0.02%
Drug: Netarsudil Ophthalmic Solution 0.04% — Topical sterile ophthalmic solution
  Arms: Netarsudil Ophthalmic Solution 0.04%
Other: Netarsudil Ophthalmic Solution Placebo — Topical sterile ophthalmic solution
  Arms: Netarsudil Ophthalmic Solution Placebo

SUMMARY:
Test ocular hypotensive efficacy and systemic safety of netarsudil 0.01%, 0.02%, 0.04% relative to placebo in subjects with open-angle glaucoma or ocular hypertension in Japan

ELIGIBILITY:
Inclusion Criteria:

1. Must be 20 years of age or older
2. Diagnosis of open-angle glaucoma (OAG) or ocular hypertension (OHT) in both eyes. (OAG in one eye and OHT in the fellow eye is acceptable)
3. BCVA 0.1 or better in decimal unit using Landolt-C chart or its equivalent
4. Able and willing to give signed informed consent and following study instructions

Exclusion Criteria:

1. Clinically significant ocular diseases
2. Pseudoexfoliation or pigment dispersion component glaucoma, history of narrow angle closure glaucoma or narrow angles
3. Previous glaucoma intraocular surgery
4. Refractive surgery in either eye
5. Ocular trauma
6. Ocular infection or inflammation
7. Known hypersensitivity to benzalkonium chloride or excipient of netarsudil ophthalmic solution
8. Cannot demonstrate proper delivery of the eye drop
9. Clinically significant abnormalities in screen lab tests
10. Clinically significant systemic disease
11. Participation in any investigational study within 30 days of screening
12. Women of child-bearing potential who are pregnant, nursing, planning a pregnancy or not using a medically acceptable form of birth control

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2019-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenji Aso, M.D., Ph.D., Study Director — Aerie Pharmaceuticals Ireland Ltd. (Japan Branch)
Locations (25):
- Japan (25):
  - Nomura Eye Clinic, Ichinomiya-shi, Aichi-ken
  - Shisui ophthalmology clinic, Shisui, Chiba
  - Nakamori Eye Clinic, Kitakyushu-shi, Fukuoka
  - Southern TOHOKU Eye Clinic, Koriyama-shi, Fukushima
  - Kusatsu Eye Clinic, Hiroshima, Hiroshima
  - Kanamori Eye Clinic, Akashi-shi, Hyōgo
  - Sameshima Eye Clinic, Kagoshima, Kagoshima-ken
  - Asahigaoka Ophthalmology, Sendai, Miyagi
  - Sugao Eye Clinic, Osaka, Osaka
  - Yubikai Kawaguchi Aozora Eye Clinic, Kawaguchi-shi, Saitama
  - Hangai Eye Institute, Saitama-shi, Saitama
  - Omiya Hamada Eye Clinic West Entrance Branch, Saitama-shi, Saitama
  - Omiya Hamada Eye Clinic, Saitama-shi, Saitama
  - Shibuya Ophthalmology Clinic, Saitama-shi, Saitama
  - Yoshimura Eye & Internal Medical Clinic, Mishima, Shiizuoka
  - Medical Corporation Muramatsu Clinic Muramatsu Eye Clinic, Susono, Shizuoka
  - Ueda Eye Clinic, Arakawa-ku, Tokyo
  - Ochanomizu Inoue Eye Clinic, Chiyoda-ku, Tokyo
  - Kiyosawa Eye Clinic, Koto-Ku, Tokyo
  - Tamagawa Eye Clinic, Ōta-ku, Tokyo
  - Seijo Clinic, Setagaya-Ku, Tokyo
  - Dogenzaka Kato Eye Clinic, Shibuya-ku, Tokyo
  - Wakabadai Eye Clinic, Shibuya-ku, Tokyo
  - Hashida Eye Clinic, Shinagawa-Ku, Tokyo
  - Watanabe Eye Clinic, Shinagawa-Ku, Tokyo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Araie M, Sugiyama K, Aso K, Kanemoto K, Kothapalli K, Kopczynski C, Senchyna M, Hollander DA. Phase 2 Randomized Clinical Study of Netarsudil Ophthalmic Solution in Japanese Patients with Primary Open-Angle Glaucoma or Ocular Hypertension. Adv Ther. 2021 Apr;38(4):1757-1775. doi: 10.1007/s12325-021-01634-9. Epub 2021 Feb 24. PMID 33629227

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 25 clinical trial sites in Japan.
Pre-assignment Details: Prior to enrollment, adult participants were to have a Screening Visit and 2 Qualification Visits to allow for washout of ocular hypotensive medication if needed.
Period: Overall Study
Arm/Group | Netarsudil Ophthalmic Solution 0.01% | Netarsudil Ophthalmic Solution 0.02% | Netarsudil Ophthalmic Solution 0.04% | Netarsudil Ophthalmic Solution Placebo
Started | 55 | 54 | 51 | 55
Completed | 54 | 53 | 46 | 54
Not Completed | 1 | 1 | 5 | 1
Not completed — Adverse Event | 1 | 1 | 4 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Netarsudil Ophthalmic Solution 0.01% | Netarsudil Ophthalmic Solution 0.02% | Netarsudil Ophthalmic Solution 0.04% | Netarsudil Ophthalmic Solution Placebo | Total
Number analyzed (Participants) | 55 | 54 | 51 | 55 | 215
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (14.62) | 64.1 (12.16) | 62 (13.56) | 64.6 (12.58) | 63.35 (13.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 29 | 27 | 31 | 123
  Male | 19 | 25 | 24 | 24 | 92
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 55 | 54 | 51 | 55 | 215
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP)
Description: Mean diurnal IOP within a treatment by Goldman Applanation Tonometry
Time Frame: 29 Days
Population: Intent to treat (ITT) population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Netarsudil Ophthalmic Solution 0.01% | Netarsudil Ophthalmic Solution 0.02% | Netarsudil Ophthalmic Solution 0.04% | Netarsudil Ophthalmic Solution Placebo
Number analyzed (Participants) | 55 | 54 | 51 | 55
mmHg
  Day 1 | 20.5 (2.8362) | 20.3 (2.8039) | 20.8 (3.2037) | 21.1 (3.7023)
  Day 8 | 16.2 (2.568) | 15.9 (2.673) | 15.7 (4.014) | 19.8 (4.059)
  Day 15 | 15.9 (2.703) | 15.6 (2.573) | 15.7 (4.190) | 19.3 (3.702)
  Day 29 | 16.3 (2.609) | 15.4 (2.411) | 16.2 (4.496) | 19.3 (3.728)
Statistical Analysis 1: Comparison: Netarsudil Ophthalmic Solution 0.01% vs Netarsudil Ophthalmic Solution 0.02% vs Netarsudil Ophthalmic Solution 0.04% vs Netarsudil Ophthalmic Solution Placebo; Test type: Superiority; p < 0.0001, ANCOVA

ADVERSE EVENTS:
Time Frame: Ocular/Systemic safety during a 4-week treatment period
Description: Safety population, defined as all randomized subjects who received at least one dose of study drug.
Arm/Group | Netarsudil Ophthalmic Solution 0.01% | Netarsudil Ophthalmic Solution 0.02% | Netarsudil Ophthalmic Solution 0.04% | Netarsudil Ophthalmic Solution Placebo
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/54 | 0/51 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/54 | 0/51 | 0/55
Other Adverse Events (participants affected / at risk) | 21/55 | 27/54 | 36/51 | 5/55
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Netarsudil Ophthalmic Solution 0.01% (N=55) | Netarsudil Ophthalmic Solution 0.02% (N=54) | Netarsudil Ophthalmic Solution 0.04% (N=51) | Netarsudil Ophthalmic Solution Placebo (N=55)
Conjunctival Hyperemia (Eye disorders) | 13 | 20 | 29 | 1
Eye Irritation (Eye disorders) | 3 | 5 | 2 | 0
Conjunctival Hemorrhage (Eye disorders) | 0 | 3 | 3 | 0
Eye Discharge (Eye disorders) | 1 | 1 | 1 | 0
Punctate keratitis (Eye disorders) | 1 | 0 | 1 | 1
Vision blurred (Eye disorders) | 1 | 1 | 1 | 0
Abnormal sensation in eye (Eye disorders) | 0 | 1 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 2 | 0
Visual acuity reduced (Eye disorders) | 0 | 1 | 1 | 0
Blepharitis (Eye disorders) | 0 | 0 | 1 | 0
Chalazion (Eye disorders) | 1 | 0 | 0 | 0
Conjunctival follicles (Eye disorders) | 0 | 0 | 1 | 0
Corneal erosion (Eye disorders) | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0
Erythema of eyelid (Eye disorders) | 1 | 0 | 0 | 0
Iritis (Eye disorders) | 0 | 0 | 1 | 0
Keratitis (Eye disorders) | 0 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 0 | 0
Retinal exudates (Eye disorders) | 0 | 0 | 1 | 0
Retinal tear (Eye disorders) | 0 | 0 | 1 | 0
Swelling of eyelid (Eye disorders) | 0 | 1 | 0 | 0
Trichiasis (Eye disorders) | 0 | 0 | 0 | 1
Ulcerative keratitis (Eye disorders) | 1 | 0 | 0 | 0
Vernal keratoconjuncitvitis (Eye disorders) | 0 | 0 | 1 | 0
Visual acuity reduced transiently (Eye disorders) | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 2 | 0 | 2 | 0
Instillation site foreign body sensation (General disorders) | 0 | 1 | 1 | 0
Instillation site pain (General disorders) | 0 | 1 | 0 | 0
Intraocular pressure increased (Investigations) | 0 | 0 | 1 | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2 | 3 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0
Gastritis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Urine leukocyte esterase positive (Investigations) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Urine abnormality (Renal and urinary disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publishing any trial results, site shall provide the to be published information to the Sponsor for review and obtain written approval at least thirty (30) days in advance of publication.

DOCUMENTS (2):
  • Study Protocol (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/45/NCT03844945/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-16): https://cdn.clinicaltrials.gov/large-docs/45/NCT03844945/SAP_001.pdf